CLINICAL TRIAL: NCT04604626
Title: Rare Obesity Cohorts With Food Behavioral Disorders : Better Diagnosis for Better Treatment
Acronym: ObeRar
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200181; 2019-A03201-56 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-04-07; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — serum, DNA, urine, stool, and adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 1: Adults and children with severe obesity ie (BMI> 35 kg / m² for adults and Z BMI score> 3DS for age and sex for children) and / or eating disorders with genetic diagnosis as part of care.
- Population 2: Adults and children with obesity and / or eating disorders hypothalamic lesion (craniopharyngioma example).

SUMMARY:
Hypothalamic obesity (HO) is defined as obesity secondary to functional or anatomical alterations of the hypothalamus, the central organ of energy homeostasis. The causes of HO are related either to hypothalamic lesions (eg craniopharyngioma) either to genetic diseases (syndromic obesity such as Prader-Willi syndrome or monogenic non syndromic obesity such as variants on leptin/melanocortin pathway). HO, which accounts for about 5 to 10% of obesity, groups complex disorders characterized by severe obesity associated with eating disorders, cognitive and behavioral disorders, endocrine and metabolic alterations and sometimes a visual deficit, with a major impact on quality of life, morbidity and mortality. There is currently no specific treatment of HO.

Clinical management is essentially behavioral, based on daily support of eating behavior and physical activities. HO is characterized by an intense and almost permanent hunger; a satiety disorder and an obsessive interest in food.

The education regarding food intake behavior of the caregivers and relateds is critical with advices concerning the control of the access to food and the setting up of a precise food frame on the quantities, with low energetic density, and schedules. HO are complex medical situations, often refractory to current lifestyle therapies. However innovative therapies with molecules targeting the hypothalamus are emerging. The investigator's main hypothesis is that HO have alterations in eating behavior that can be improved by innovative treatments such as, for example, molecule targeting the melanocortin pathway. The response to therapy could depend on hypothalamic origin and especially on the genotype. ObeRar cohort aims to i) improve early diagnosis of HO and ii) characterize the natural history of obesity and eating disorders, the associated phenotypes and "lifestyle" profiles (physical activity, sleep, nutrition) and cardio-metabolic and neuropsychological parameters. Defining profiles will help personalize individual care management and target patients who can participate in clinical trials with innovative therapeutics. ObeRar-cohort will thus improve the early diagnosis, prognosis, medical management and innovative therapies of these particularly severe forms of rare obesities.

DETAILED DESCRIPTION:
Hypothalamic obesity (HO) is defined as a rare obesity secondary to impaired functioning of the hypothalamus nuclei, the central organ of energy and weight homeostasis. Among the causes of HO, there are those related to a hypothalamic lesion (lesional) such as craniopharyngioma (CP) or inflammatory (sarcoidosis, tuberculosis etc ..) and those called genetic, with variations in gene involved in the central regulation of energy homeostasis. The genetic causes of obesity can be either "monogenic" by mutation of genes involved in the leptin / melanocortin pathway, or "syndromic", defined by the association of obesity and other clinical signs (syndrome), especially neuropsychological traits, such as Prader-Willi syndrome (PWS) or Bardet-Biedl syndrome. PWS, which has a frequency of 1/15000 births, is one of the most well-known obesity-related syndromes. PWS is characterized by muscle hypotonia at birth, severe hyperphagia and food impulsivity, dysmorphic features, and intellectual disability with cognitive-behavioral abnormalities. Monogenic obesity involves rare clinical situations with variants in one of the genes in the MC4R pathway, which plays a pivotal role in the hypothalamic control of food intake and energy expenditure. To date, at least 10 genes directly involved in or regulating the leptin/melanocortin pathway are known: leptin (LEP), leptin receptor (LEPR), pro-opiomelanocortin (POMC), prohormone convertase 1 (PCSK1), melanocortin receptor type 4 (MC4R) and its regulator Melanocortin Receptor Accessory Protein 2 (MRAP2), single -minded homolog 1 (SIM1), brain-derived neurotrophic factor (BDNF), neurotrophic tyrosine kinase receptor type 2 (NTRK2) and more recently, adenylate cyclase 3 (ADCY3). It is of interest to mention that some genes involved in syndromic obesity, such as PWS and BBS, are also involved in the MC4R pathway.

Although HO has various pathophysiological origins, there are common linked phenotypes with the presence of severe obesity and abnormal food intake behovior, having a heavy impact on the morbidity and mortality. Obesity is multifactorial, associated with an increase in energy intake, a decrease in energy expenditure and an alteration of peripheral metabolism with abnormal organ cross-talks. People with HO have often cognitive deficits, learning difficulties and social skills disorders. These factors alter patients' quality of life. At present, there is no specific treatment of HO. Drug treatments have been proposed such as melatonin, somatostatin analogue or sympathomimetics but with limited effects on weight and feeding behavior, resulting in no prescribing recommendations given the lack of randomized studies with sufficient patient samples. Sibutramine tested in patients with lesional or genetic HO was withdrawed from the market in France since 2010 for potentially deleterious effects on the cardiovascular system. GLP 1 analogues are an interesting therapeutic approach in patients with craniopharyngioma with some efficacy on weight, but are currently dedicated for diabetic patients in France. Regarding bariatric surgery in rare and secondary obesities, the French Haute Autorité de Santé recommends that "the indication must be exceptional and discussed on a case by case basis".

So current management is essentially behavioral, based on daily support of eating behavior and physical activity. Food management requires from a very young age and during the whole life, a permanent food control, to fight against primary impulsivity of central origin, can be a cause of frustration and behavioral disorders. Indeed, the hypothalamic impairment is characterized by intense and permanent hunger, a lack of satiety and an obsession for food. The affected patients are completely overwhelmed by this addictive behavior. It is extremely difficult or impossible for the child as for the adult with this syndrome to control his dietary intake. The caregivers and relateds must therefore control access to food at home and abroad. This requires constant supervision. An early education of food in the family is essential because today it there is no possible and sustainable autonomy regarding diet for these patients.

So, if the global, specialized and multidisciplinary care is to be implemented as early as possible, from early childhood, the development of new therapeutic strategies is essential due to the severe and early obesity. In recent years, research in therapeutic innovation has developed in an interesting way in genetic obesity, in particular by targeting the melanocortin pathway. HO have various origins but have a common phenotype, that is the presence of eating disorders with hyperphagia and food impulsivity. This is responsible for weight gain which can lead to obesity, having a significant impact on the morbidity and mortality. However, no precise data are available currently on the specific phenotype of each origin, the genotype/phenotype correlation, and national medical history of OH throughout life, from birth to adulthood, as well as the associated phenotypes, are still to be precisely described.

ELIGIBILITY:
Inclusion Criteria:

* Population 1:

  1. Adults ≥ 18 years old with BMI> 35 kg / m² or children <18 years old with BMI Zscore> + 3DS for age and sex and / or eating behavior disorders consulting in one of the participating centers
  2. Patient benefiting from a genetic diagnosis as part of his usual care according to criteria justifying a genetic analysis such as:

     obesity with early onset (<12 years) or very severe BMI> 50 kg / m² and / or presence of eating disorders, endocrine abnormalities or other symptoms suggestive of a genetic anomaly (such as: intellectual disability, retinopathy of pigmentation or other)
  3. Adult patient or holders of parental authority (for children) having received the information and having signed a free, informed and written consent (or for adult patients under legal protection measure or unable to consent, information and obtaining the consent of the legal representative, the support person, or the relative / close relative).
* Population 2

  1. Adult or child with obesity and / or eating disorder due to hypothalamic lesion (craniopharyngioma for example)
  2. Adult patient or holders of parental authority (for children) having received the information and having signed a free, informed and written consent (or for adult patients under legal protection measure or unable to consent, information and obtaining the consent of the legal representative, the support person, the relative / relative).

Exclusion Criteria:

1. Refusing to participate in the study
2. Not mastering the french language
3. Safety measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population 1: Adults and children with severe obesity ie (BMI> 35 kg / m² for adults and Z BMI score> 3DS for age and sex for children) and / or eating disorders with genetic diagnosis as part of care This population will be divided into 5 groups according to the genetic diagnosis made
  * Prader willi syndrome (SPW)
  * syndromic obesity except prader willi (OS)
  * obesity by homozygous mutation of the melanocortin pathway (HomMel)
  * obesity by heterozygous mutation of the melanocortin pathway (HetMel)
  * controls without genetic abnormality found in view of the final results of the genetic diagnosis(CON) Population 2: Adults and children with obesity and / or eating disorders hypothalamic lesion (craniopharyngioma example)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2040-07-01 (Estimated)

PRIMARY OUTCOMES:
This criterion is the age of obesity beginning | For adults, at inclusion. For children at inclusion and every three years (from date of inclusion until the date of first documented BMI>IOTF 30 kg/m²) (e.g from date of inclusion until the end of follow up, so 20 years)
  A BMI curve is performed using the aggregation of multiple measurements (eg weight in kg and height in meters) during childhood. Retrospective data on height and weight collected every year form birth to the age BMI= weight/height², Obesity is defined for a BMI above the IOTF curve

SECONDARY OUTCOMES:
Maximum weight in kg | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  allows to define the severity of obesity
Maximum height in m | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  allows to calculate the maximum BMI= maximum weight/(maximum height)²
Adult: number of calories/24h with distribution of macronutrients | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  from the dietary survey costed by a dietician with kcal/24h and repartition of % of glucids, lipids and proteins
Adult: binge eating behavior | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Binge eating scale (BES) (score 0-30, a score > 18 defines the presence of hyperphagia)
Adult: hyperphagia | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Dyckens hyperphagia questionnaire for entourage if the patient is not unable to complete questionnaires due to intellectual or other disabilities (a score>9 is considered as the limit for hyperphagia)
Adult: hunger and satiety before and after meals | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Score on the visual analogic scale (VAS) (min 0-max 10, a score >6 is considered as high)
Adult: Quantification of physical activity in minutes / day | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  count of mouvements/day measured by an accelerometer
Adult: waist circumference | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  a wais curcumeference greater than 102 cm (in men or greater than 88 cm ) in women is the current threshold for increased metabolic risk (caucasian population)
Adult: percentage of fat mass | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  DEXA
Adult: quantification of visceral fat in cm² | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  scan
Adult: Quality of life | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  the The Short Form (36) Health Survey (SF36) is as standardized questionnaire to assess quality of life. The SF-36 yields eight scale scores and two summary scores: the physical component summary (PCS) and mental component summary (MCS) scores
Adult: depression and anxiety | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Hospital Anxiety and depression scale (HAD) is a questionnaire with 14 questions with a score of anxiety and a score of depression (min 0-max 21)
Adult: Resting energy expenditure | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  by indirect calorimetry in kcal / 24h
Adult: Metabolic assessment | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  this complete metabolic assessment include blood measurment of routine biomarkers : total cholesterol HDLC/LDLC triglycerid glycemia in mmol/l ; insulinemia in µU/ml ; ASAT/ALAT/ gammaGT in UI/l If at least one of this marker is above the normal range, we consider that metabolic assessment is abnormal
Adult: ejection fraction | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  measurements made during cardiac MRI
Adult: Total Intelligence quotient | at the inclusion
  measured during the neuropsychological assessment if applicable (patient with intellectual disability) by the WAIS-IV tool , intellectual deficiency is considered if total IQ<70
Adult: Assessment of interoceptive capacities: counting of heartbeats | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  according to validated technique (Schandry 1981) associated with metacognitive confidence measures in the counting of heartbeats (after each answer: "how confident are you in your answer"), an auto-questionnaire of interception: MAIA (translation by T Similowsky, validated by Carré 2014) an auto-questionnaire of interception: MAIA (translation by T Similowsky, validated by Carré 2014)
Adult: Family history of obesity (parents, siblings) | at inclusion and during follow-up evaluation visit every 5 years (e.g from date of inclusion until the end of follow up, so 20 years)
  maximal BMI (Body Mass index) of mother, father, sisters and brothers
Children: Age of adiposity rebound (years) determined | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  on the BMI curve
Children: Severity of obesity | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  BMI Zscore by age and sex
Children: number of calories and distribution of macronutrients | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  from the dietary survey costed by a dietician with kcal/24h and repartition of % of glucids, lipids and proteins
Children: hunger and satiety before and after meals | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Score on the visual analogic scale (VAS) (min 0-max 10, a score >6 is considered as high)
Children: Quantification of physical activity in min / day | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  count of mouvements/day measured by an accelerometer
Children: waist circumference | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  a waist circumference greater than 102 cm (in men or greater than 88 cm ) in women is the current threshold for increased metabolic risk (caucasian population)
Children: percentage of fat mass | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  DEXA
Children: Resting energy expenditure | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  by indirect calorimetry in kcal / 24h
Children: lipids, HOMA-IR, liver enzymes | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  complete metabolic assessment
Children: IGF1, FT4, TSH, testosterone, vitamin D, PTH, others according to the clinical picture | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Complete endocrine assessment
Children: ejection fraction | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  measurement with heart ultrasound
Children: Total Intelligence quotient | at the inclusion
  measured during the neuropsychological assessment if applicable (patient with intellectual disability) by the WAIS-IV tool , intellectual deficiency is considered if total IQ<70
Children: Quality of life | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  SF10 completed by parents or SF36 by children over 15 years
Children: Hyperphagia | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Dyckens hyperphagia questionnaire completed by parents. (a score>9 is considered as the limit for hyperphagia)
Children: Food behaviour | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  questionnaire depends on the age: (0-23 months) BEBQ (Baby Eating Behavior Questionnaire) completed by parents; (2-15 years) CEBQ (Child Eating Behaviour Questionnaire) completed by parents; TFEQ21 score completed by children ( for Children >15years)
Children : over 15 years old : binge eating behavior | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Binge eating scale (BES) (score 0-30, a score > 18 defines the presence of hyperphagia)
Children : over 15 years old : depression and anxiety | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Hospital Anxiety and depression scale (HAD) is a questionnaire with 14 questions with a score of anxiety and a score of depression (min 0-max 21)
Children : over 15 years old : addiction | at inclusion and during follow-up evaluation visit every 3 years (e.g from date of inclusion until the end of follow up, so 20 years)
  Yale Food Addiction Scale (YFAS) is a 25-point questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTINE POITOU-BERNERT, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, AP-HP -Nutrition department, La Defense, France